CLINICAL TRIAL: NCT07082634
Title: Evaluation of Immediate Implant Placement Using the Socket Shield Technique in Maxillary Esthetic Zone (Clinical and Radiographic Study)
Brief Title: Immediate Implant Placement Using the Socket Shield Technique in Maxillary Esthetic Zone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-H-0176-D-M-0796
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Socket Shield Technique; Maxillary Esthetic Zone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Socket shield and immediate implant (Experimental)
  Interventions: Procedure: Socket shield concept and immediate implant placement

INTERVENTIONS:
Procedure: Socket shield concept and immediate implant placement — Tooth Sectioning: The tooth will be sectioned mesiodistally using a fissure bur, preserving the buccal segment.
  Palatal fragment extraction: carefully after sectioning the tooth , the palatal fragment is luxated and extracted with the most important factor is taking care of the buccal part not to become loose , the extraction is done using a periotome to be minimally invasive and to preserve the bone from major damage.
  Shield Preparation: The buccal fragment is reduced to bone level using a round bur, a beveled edge is created using a diamond football bur, and the shield is thinned to maintain structural integrity.
  Implant Site Preparation: Sequential osteotomy performed under copious irrigation, ensuring primary stability.
  Implant Placement: A Megagen implant is inserted

SUMMARY:
Immediate implant placement in the esthetic zone is an approach that helps preserve soft and hard tissue architecture. However, post extraction bone resorption is still a significant challenge. The socket shield technique (SST) has emerged as a promising way for preserving the buccal plate, potentially improving implant stability and reducing radiographic bone loss. The aim of the present study is to evaluate the clinical and radiographic outcomes of the socket shield technique in the maxillary esthetic zone by assessing implant stability, radiographic bone loss as well as esthetic outcome over a specified follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a non-restorable maxillary tooth in the aesthetic zone indicated for extraction and subsequent immediate implant placement.
* Patients with extraction socket Type I.
* A good standard of oral hygiene.

Exclusion Criteria:

* Patients with extraction socket Type II or III, with defect in the buccal plate.
* Absence of at least 2 mm bone apical to the extraction socket, necessary to obtain adequate primary stability for the implant assessed by pre-operative radiographic evaluation.
* The presence of any local factor that may interfere with extraction as tooth ankylosis.
* Patients with deciduous teeth.
* Patients with bruxism
* Heavy smokers.
* Systemic conditions that are considered as a contraindication for placement of implant or those that may interfere with wound healing and immunocompromised conditions and uncontrolled autoimmune diseases.
* History of oral or intravenous bisphosphonate therapy or any treatments with other medications that may interfere with bone metabolism within the past 12 months.
* Patients receiving radiotherapy or chemotheraphy.
* Patient with active infection or chronic infection with severe bone loss.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | baseline, 7, 14, and 21 days
  Pain will be evaluated, using visual analogue scale (VAS) as follows:
  (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe) (Figure 1)
Change in implant stability | baseline and 6 months
  The base line primary Implant Stability Quotient (ISQ) will be measured at the time of implant placement, while the secondary stability quotient will be measured after 6months during the prosthetic phase preparation.

SECONDARY OUTCOMES:
Change in post operative healing | baseline, 7, 14, and 21 days
  The wound healing will be assessed based on Landry Wound Healing Index. The Landry Index uses a numerical score based on the assessment of four given parameters (Erythema., Edema, Wound Margin Adaptation, and Presence of Exudate). Each parameter is given a score depending on its severity, and the total score determine an overall evaluation of wound healing
change in crestal alveolar process width | baseline and 6 months
  The width of the crestal alveolar process will be assessed by determination of the dimensional changes of Bucco-palatal ridge in the 6 months' scan. Measurements will be taken from the preoperative records and compared to those taken in the 6 month ones.
change in labial bone thickness | baseline and 6 months
  the assessment of the thickness labial plate of bone in the scan performed after 6 months and comparing it with the preoperative CBCT scans.

CONTACTS AND LOCATIONS:
Locations (1):
- Beirut Arab University, Beirut, Lebanon